CLINICAL TRIAL: NCT00942968
Title: FRAG-A001-401: Dalteparin Sodium Injection (Fragmin), Multicenter, Open-Label, Single-arm, Long Term (52 Weeks) Study for Understanding the Safety and Efficacy in Subjects With Malignancies and Symptomatic Venous Thromboembolism
Brief Title: Evaluation of Dalteparin for Long-term (One Year) Treatment of Blood Clots in Subjects With Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRAG-A001-401; A6301095 (Other: Alias Study Number)
Record Dates: First submitted 2009-07-16; First posted 2009-07-21 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: dalteparin

INTERVENTIONS:
Drug: dalteparin — Daily subcutaneous injection 200IU/kg dalteparin

SUMMARY:
The purpose of this study is to determine the long term tolerability and safety of dalteparin in subjects with cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, age greater than or equal to 18 years of age.
2. Females should be either of non-childbearing potential as a result of surgery, radiation therapy, menopause (one year post onset), or of childbearing potential and willing to adhere to an acceptable method of pregnancy prevention.
3. Subjects must be newly diagnosed, symptomatic proximal deep-vein thrombosis of the lower extremity, pulmonary embolism, or both.
4. Subjects must have active malignancy defined as a diagnosis of cancer (excluding basal cell or squamous cell carcinoma of the skin) within six months before enrollment, having received any treatment for cancer within the previous six months, or having documented recurrent or metastatic cancer.
5. Prior to enrollment, subjects must not have received therapeutic doses of anticoagulant therapy (including low molecular weight heparin [LMWH]) for >48 hours (or >4 doses within 48 hours).
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
7. Subjects must have a life expectancy of >6 months.
8. Subjects must have a platelet count of >75,000 mm^3.
9. The subject must not be on any oral anticoagulant therapy for concomitant diseases.
10. Subjects must have no active or serious bleeding episodes within two weeks prior to study entry.
11. Subjects must be able to comply with scheduled follow-ups.

Exclusion Criteria:

1. Subjects who have a high risk of serious bleeding (e.g., recent neurosurgery within 30 days, history of intracranial hemorrhage, acute gastroduodenal ulcer, etc.).
2. Subjects who are on hemodialysis.
3. Subjects who have a prior placement of a Greenfield filter or other device to prevent embolization of deep vein thromboses.
4. Subjects with a known contraindication to the use of heparin (e.g., heparin-induced thrombocytopenia).
5. Subjects with a known hypersensitivity to heparin, dalteparin sodium, other LMWHs or pork products.
6. Subjects who are currently participating in another clinical trial involving anticoagulation therapy (with the exception of acetylsalicylic acid (ASA) in the 30 days prior to study entry, or who are actively using any investigational drugs/treatments 30 days prior to study entry involving anticoagulation therapy (with the exception of ASA , t.i.d).
7. Subject is pregnant or breast feeding.
8. Subjects with uncontrolled hypertension characterized by a sustained systolic pressure >170 mmHg and/or diastolic pressure >100 mmHg.
9. Subjects with a serious concomitant systemic disorder (for example, active infection including HIV or cardiac disease) that in the opinion of the investigator, would compromise the subject's ability to complete the study.
10. Any condition that makes the subject unsuitable in the opinion of the investigator.
11. Subjects with leukemia or myeloproliferative syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2009-06; Primary Completion 2012-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Gary Palmer, MD, Study Director — Medical Affairs, Eisai, Inc
Locations (42):
- United States (21):
  - Arizona Cancer Center, Tucson, Arizona
  - Bay Area Cancer Research Group, Pleasant Hill, California
  - Harbor-UCLA Medical Center, Torrance, California
  - University of CT Health Center, Farmington, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Georgetown University Hospital-Lombardi Cancer Ctr, Washington D.C., District of Columbia
  - Halifax Health, Daytona Beach, Florida
  - Atlanta Institute for Medical Research, Decatur, Georgia
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Bringham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital K-15, Detroit, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University, Medical Center, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - MidDakota Clinic, Bismarck, North Dakota
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Vermont Cancer Center at Fletcher Allen Health Care, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
- Austria (6):
  - LKH Graz Univrsitatstklinik fur Innere Medizin, Graz
  - Medizinische Universitat Innsbruck Studienambulanz Hamatologie, Innsbruck
  - KH d. Elizabethinen Linz GmbH Servicestelle fur klin. Studien und Universitare Angelegenheiten, Linz
  - KH der Barmherzigen Schwestern, Linz
  - Dialysestation Landesklinkum St.Poelten, Sankt Pölten
  - Medizinische Universitat Wien, Vienna
- Canada (8):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Ottawa Health Research Institute, Ottawa, Ontario
  - University Health Network-Toronto General Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
- Netherlands (2):
  - Gelre Ziekenhuizen-Locatie Apeldoorn, Apeldoorn
  - Orbis Medisch Centrum, Sittard-Geleen, Sittard-Geleen
- Spain (5):
  - Hospital clinic i Provincial de Agencia de Ensayos Clinicos, Barcelona
  - Hospital General Santa Maria del Rosell, Caragena (Murcia)
  - Hospital Virgen de la Arrixaca, El Palmar (Murcia)
  - Hospital Universitari Dr Josep Trueta, Girona
  - Clinica Universitaria de Navarra, Pamplona

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=FRAG-A001-401&StudyName=Daleparin%20Sodium%20Injection%20%28fragmin%20%28registered%29%29%2C%20Multicenter%2C%20Open%20Label%2C%20Single-arm%2C%20Long%20Term%20%2852%20Weeks%29%20Study%20For%20Underatnding%20Safety%20And%20Efficacy%20In%20Subjects%20With%20Malignancies%20And%20Symptomatic%20Venous%20Thromboembolism

RESULTS

PARTICIPANT FLOW:
Groups:
- Dalteparin Sodium: Participants received subcutaneous (SC) injection of dalteparin sodium 200 international units per kilogram (IU/kg) once daily (QD) from Week 1-4 followed by SC injection of dalteparin sodium 150 IU/kg QD from Week 5-52.
Period: Overall Study
Arm/Group | Dalteparin Sodium
Started | 338
Treated | 334
Completed | 109
Not Completed | 229
Not completed — Adverse Event | 60
Not completed — Death | 76
Not completed — Protocol Violation | 9
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 44
Not completed — Sponsor request | 5
Not completed — Physician Decision | 11
Not completed — Progression of disease | 12
Not completed — Inferior vena cava filter placement | 4
Not completed — Pulmonary embolism (PE) | 1
Not completed — Participant required pancreatic biopsy | 1
Not completed — Deep vein thrombosis (DVT) | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 treatment with dalteparin sodium.
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171
  Male | 163

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Bleeding Events Adjudicated by Central Adjudication Committee
Description: A bleeding event was considered as major if it was clinically overt and satisfies 1 or more of the following criteria: 1) bleeding accompanied by a decrease in hemoglobin of greater than or equal to (>=) 2 gram per deciliter (g/dL), 2) bleeding occurred at a critical site (intraocular, spinal/epidural, intracranial, retroperitoneal, or pericardial bleeding), 3) bleeding leads to a transfusion of two or more units of packed red blood cells, 4) bleeding leads to death. In this outcome measure, number of participants with major bleeding events (adjudicated by Central Adjudication Committee) were reported.
Time Frame: Month 2 up to Month 6
Population: Safety population included all participants who received at least 1 treatment with dalteparin sodium.
Measure: Number; unit: participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
participants | 14

2. Primary Outcome: Number of Participants With Major Bleeding Events Adjudicated by Central Adjudication Committee
Description: A bleeding event was considered as major if it was clinically overt and satisfies 1 or more of the following criteria: 1) bleeding accompanied by a decrease in hemoglobin of >=2 g/dL, 2) bleeding occurred at a critical site (intraocular, spinal/epidural, intracranial, retroperitoneal, or pericardial bleeding), 3) bleeding leads to a transfusion of two or more units of packed red blood cells, 4) bleeding leads to death. In this outcome measure, number of participants with major bleeding events (adjudicated by Central Adjudication Committee) were reported.
Time Frame: Month 7 up to Month 12
Population: Safety population included all participants who received at least one 1 treatment with dalteparin sodium.
Measure: Number; unit: participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
participants | 8

3. Primary Outcome: Number of Participants With New or Recurrent Venous Thromboembolism (VTE) Adjudicated by Central Adjudication Committee
Description: VTEs included both deep vein thrombosis (DVT) and pulmonary embolism (PE). DVT is a blood clot in the deep veins of the leg. If a DVT clot breaks off (embolizes) from a vein wall and flows towards the lungs and blocks some or all of the blood supply, it becomes pulmonary embolism (PE). When a blood clot (thrombus) breaks, loose and travels in the blood, this is called a venous thromboembolism. DVT was diagnosed using either computed tomography scan or contrast venography. PE was diagnosed by either radionuclide ventilation-perfusion studies, contrast CT scan or an angiogram. In this outcome measure, number of participants with new or recurrent VTE (adjudicated by Central Adjudication Committee) were reported.
Time Frame: Month 7 up to Month 12
Population: Efficacy analysis population included all participants who received at least 1 study treatment with dalteparin sodium. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 194
participants | 8

4. Secondary Outcome: Number of Participants With Investigator Identified Major Bleeding Events
Description: A bleeding event was considered as major if it was clinically overt and satisfies 1 or more of the following criteria: 1) bleeding accompanied by a decrease in hemoglobin of >=2 g/dL, 2) bleeding occurred at a critical site (intraocular, spinal/epidural, intracranial, retroperitoneal, or pericardial bleeding), 3) bleeding leads to a transfusion of two or more units of packed red blood cells, 4) bleeding leads to death. In this outcome measure, number of participants with major bleeding events (identified by investigator) were reported.
Time Frame: Month 1 up to Month 6; Month 7 up to Month 12; Month 1 up to Month 12; Month 2 up to Month 6; Month 2 up to Month 12
Population: Safety population included all participants who received at least 1 treatment with dalteparin sodium.
Measure: Number; unit: participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
participants
  Month 1 up to Month 6 | 28
  Month 7 up to Month 12 | 7
  Month 1 up to Month 12 | 35
  Month 2 up to Month 6 | 15
  Month 2 up to Month 12 | 22

5. Secondary Outcome: Number of Participants With Any Bleeding Event (Major or Minor) Adjudicated by Central Adjudication Committee
Description: A bleeding event was considered as major if it was clinically overt and satisfies 1 or more of the following criteria: 1) bleeding accompanied by a decrease in hemoglobin of >=2 g/dL, 2) bleeding occurred at a critical site (intraocular, spinal/epidural, intracranial, retroperitoneal, or pericardial bleeding), 3) bleeding leads to a transfusion of two or more units of packed red blood cells, 4) bleeding leads to death. A bleeding event was considered as minor if it was clinically overt but not meeting the criteria for major bleeding. In this outcome measure, number of participants with any (major or minor) bleeding events (adjudicated by Central Adjudication Committee) were reported.
Time Frame: Month 1 up to Month 6, Month 7 up to Month 12, Month 1 up to Month 12, Month 2 up to Month 6, and Month 2 up to Month 12
Population: Safety population included all participants who received at least 1 treatment with dalteparin sodium.
Measure: Number; unit: participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
participants
  Month 1 up to Month 6 | 91
  Month 7 up to Month 12 | 21
  Month 1 up to Month 12 | 112
  Month 2 up to Month 6 | 47
  Month 2 up to Month 12 | 68

6. Secondary Outcome: Number of Participants With Fatal Bleeding Events
Description: Fatal bleeding events refers to those bleeding events which leads to death of participant. In this outcome measure, number of participants with fatal bleeding events were reported.
Time Frame: Month 1 up to Month 6; Month 7 up to Month 12; Month 1 up to Month 12; Month 2 up to Month 6; Month 2 up to Month 12
Population: Safety population included all participants who received at least 1 treatment with dalteparin sodium.
Measure: Number; unit: participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
participants
  Month 1 up to Month 6 | 1
  Month 7 up to Month 12 | 1
  Month 1 up to Month 12 | 2
  Month 2 up to Month 6 | 1
  Month 2 up to Month 12 | 2

7. Secondary Outcome: Time to First Occurrence of Major Bleeding Event Adjudicated by Central Adjudication Committee
Description: Time to first occurrence of major bleeding event was defined as the time interval (in days) between the date of first study treatment and the date of documentation of first major bleeding event. A bleeding event was considered as major if it was clinically overt and satisfies 1 or more of the following criteria: 1) bleeding accompanied by a decrease in hemoglobin of >=2 g/dL, 2) bleeding occurred at a critical site (intraocular, spinal/epidural, intracranial, retroperitoneal, or pericardial bleeding), 3) bleeding leads to a transfusion of two or more units of packed red blood cells, 4) bleeding leads to death.
Time Frame: Month 1 up to Month 12
Population: Safety population included all participants who received at least 1 treatment with dalteparin sodium.
Measure: Mean (Standard Error); unit: days
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
days | 332.9 (5.25)

8. Secondary Outcome: Time to First Occurrence of Any Bleeding Event (Major or Minor) Adjudicated by Central Adjudication Committee
Description: Time to first occurrence of any bleeding event was defined as the time interval (in days) between the date of first study treatment and the date of documentation of first bleeding event (major or minor). A bleeding event was considered as major if it was clinically overt and satisfies 1 or more of the following criteria: 1) bleeding accompanied by a decrease in hemoglobin of >=2 g/dL, 2) bleeding occurred at a critical site (intraocular, spinal/epidural, intracranial, retroperitoneal, or pericardial bleeding), 3) bleeding leads to a transfusion of two or more units of packed red blood cells, 4) bleeding leads to death. A bleeding event was considered as minor if it was clinically overt but not meeting the criteria for major bleeding.
Time Frame: Month 1 up to Month 12
Population: Safety population included all participants who received at least 1 treatment with dalteparin sodium.
Measure: Mean (Standard Error); unit: days
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
days | 262.5 (8.52)

9. Secondary Outcome: Number of Participants With Investigator Identified New or Recurrent Venous Thromboembolism (VTEs)
Description: VTEs included both DVT and PE. DVT is a blood clot in the deep veins of the leg. If a DVT clot breaks off (embolizes) from a vein wall and flows towards the lungs and blocks some or all of the blood supply, it becomes PE. When a blood clot (thrombus) breaks, loose and travels in the blood, this is called a venous thromboembolism. DVT was diagnosed using either computed tomography scan or contrast venography. PE was diagnosed by either radionuclide ventilation-perfusion studies, contrast CT scan or an angiogram. In this outcome measure, number of participants with new or recurrent VTE (identified by investigator) were reported.
Time Frame: Month 1 up to Month 6; Month 7 up to Month 12; Month 1 up to Month 12; Month 2 up to Month 6; Month 2 up to Month 12
Population: Efficacy analysis population included all participants who received at least 1 study treatment with dalteparin sodium. Here, 'n' signifies those participants who were evaluable at specified time intervals.
Measure: Number; unit: participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
participants
  Month 1 up to Month 6 (n=334) | 29
  Month 7 up to Month 12 (n=195) | 8
  Month 1 up to Month 12 (n=334) | 37
  Month 2 up to Month 6 (n=295) | 9
  Month 2 up to Month 12 (n=295) | 17

10. Secondary Outcome: Number of Participants With New or Recurrent Venous Thromboembolism (VTE) or Central Venous Thrombosis (CVT) Adjudicated by Central Adjudication Committee
Description: VTEs included both DVT and PE. DVT is a blood clot in the deep veins of the leg. If a DVT clot breaks off (embolizes) from a vein wall and flows towards the lungs and blocks some or all of the blood supply, it becomes PE. When a blood clot (thrombus) breaks, loose and travels in the blood, this is called a venous thromboembolism. DVT was diagnosed using either computed tomography scan or contrast venography. PE was diagnosed by either radionuclide ventilation-perfusion studies, contrast CT scan or an angiogram. CVT is blood clot of the venous channels in the brain. CVT was diagnosed by contrast venography or ultrasonography. In this outcome measure, number of participants with new or recurrent VTE or CVT (adjudicated by Central Adjudication Committee) were reported.
Time Frame: Month 1 up to Month 6; Month 7 up to Month 12; Month 1 up to Month 12; Month 2 up to Month 6; Month 2 up to Month 12
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
participants
  Month 1 up to Month 6 (n=334) | 29
  Month 7 up to Month 12 (n=194) | 8
  Month 1 up to Month 12 (n=334) | 37
  Month 2 up to Month 6 (n=296) | 10
  Month 2 up to Month 12 (n=296) | 18

11. Secondary Outcome: Number of Participants With Investigator Identified New or Recurrent Venous Thromboembolism (VTE) or Central Venous Thrombosis (CVT)
Description: VTEs included both DVT and PE. DVT is a blood clot in the deep veins of the leg. If a DVT clot breaks off (embolizes) from a vein wall and flows towards the lungs and blocks some or all of the blood supply, it becomes PE. When a blood clot (thrombus) breaks, loose and travels in the blood, this is called a venous thromboembolism. DVT was diagnosed using either computed tomography scan or contrast venography. PE was diagnosed by either radionuclide ventilation-perfusion studies, contrast CT scan or an angiogram. CVT is blood clot of the venous channels in the brain. CVT was diagnosed by contrast venography or ultrasonography. In this outcome measure, number of participants with new or recurrent VTE or CVT (identified by investigator) were reported.
Time Frame: Month 1 up to Month 6; Month 7 up to Month 12; Month 1 up to Month 12; Month 2 up to Month 6; Month 2 up to Month 12
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
participants
  Month 1 up to Month 6 (n=334) | 29
  Month 7 up to Month 12 (n=195) | 8
  Month 1 up to Month 12 (n=334) | 37
  Month 2 up to Month 6 (n=295) | 9
  Month 2 up to Month 12 (n=295) | 17

12. Secondary Outcome: Time to First Occurrence of New or Recurrent Venous Thromboembolism (VTE) Adjudicated by Central Adjudication Committee
Description: Time to first occurrence of new or recurrent VTE was defined as the time interval (in days) between the date of first study treatment and the date of documentation of first VTE. VTEs included both DVT and PE. DVT is a blood clot in the deep veins of the leg. If a DVT clot breaks off (embolizes) from a vein wall and flows towards the lungs and blocks some or all of the blood supply, it becomes PE. When a blood clot (thrombus) breaks, loose and travels in the blood, this is called a venous thromboembolism. DVT was diagnosed using either computed tomography scan or contrast venography. PE was diagnosed by either radionuclide ventilation-perfusion studies, contrast CT scan or an angiogram.
Time Frame: Month 1 up to Month 12
Population: Efficacy analysis population included all participants who received at least 1 study treatment with dalteparin sodium.
Measure: Mean (Standard Error); unit: days
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
days | 294.1 (4.87)

13. Secondary Outcome: Time to First Occurrence of New or Recurrent VTE or CVT Adjudicated by Central Adjudication Committee
Description: Time to first occurrence of new or recurrent VTE or CVT was defined as the time interval (in days) between the date of first study treatment and the date of documentation of first VTE or CVT. VTEs included both deep vein thrombosis (DVT) and pulmonary embolism (PE) .DVT is a blood clot in the deep veins of the leg. If a DVT clot that breaks off (embolizes) from a vein wall and flows towards the lungs and blocks some or all of the blood supply, it becomes pulmonary embolism (PE). When a blood clot (thrombus) breaks, loose and travels in the blood, this is called a venous thromboembolism. DVT was diagnosed using either computed tomography scan, contrast venography or contrast venography. PE was diagnosed by either radionuclide ventilation-perfusion studies, contrast CT scan or an angiogram. CVT is blood clot of the venous channels in the brain. CVT was diagnosed by contrast venography or ultrasonography.
Time Frame: Month 1 up to Month 12
Population: Efficacy analysis population included all participants who received at least 1 study treatment with dalteparin sodium.
Measure: Mean (Standard Error); unit: days
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
days | 294.1 (4.87)

14. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Week 52 that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline (Day 1) up to Week 52
Population: Safety population included all participants who received at least 1 treatment with dalteparin sodium.
Measure: Number; unit: participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
participants
  AE | 328
  SAE | 213

15. Other Pre Specified Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Criteria for abnormality: Hemoglobin greater than or equal to(>=)130*lower limit of normal(LLN); less than or equal to(<=)170*upper limit of normal(ULN), hematocrit >=0.39*LLN;<=0.51*ULN, red blood cell >=4.5*LLN;<=5.9*ULN, platelet>=150*LLN;<= 450*ULN, white blood cells >=4*LLN;<=11*ULN; lymphocytes>=0.09;<=0.44, neutrophils=>0.16*LLN;<=0.7*ULN, eosinophils<=0.04*ULN, basophils<=0.02*ULN, monocytes>0.08*ULN; bilirubin >=5.1*LLN;<=22.2*ULN, aspartate aminotransferase >=13*LLN;<=36*ULN, alanine aminotransferase>=11*LLN;<=54*ULN, alkaline phosphatase>=31*LLN ;<=104 *ULN, total protein>=60*LLN; <=76*ULN, albumin=>35*LLN;<=50*ULN, glucose>=3.77 ;<=6.05;blood urea nitrogen>=1.785*LLN;<=7.5*ULN, creatinine>=70.7*LLN;<=114.9*ULN, creatinine kinase>=30*LLN ;<=280*ULN, lactate dehydrogenase>=85*LLN;<=180*ULN, sodium>=137*LLN ;<=144*ULN, potassium >=3.5*LLN;<=5*ULN, chloride>=102*LLN;<=111*ULN, calcium>=2.22*LLN ;<=2.57*ULN, phosphorus=>0.81 ;<=1.45); nitrogen cholesterol>=1.78*LLN ;<=7.49*ULN.
Time Frame: Baseline (Day 1) up to Week 52
Population: Safety population included all participants who received at least 1 treatment with dalteparin sodium.
Measure: Number; unit: participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
participants | 0

16. Other Pre Specified Outcome: Number of Participants With Abnormal Physical Examinations Findings
Description: Physical examinations included head, ears, nose, throat (ENT), neck, heart, chest, lungs, abdomen, extremities, neurological systems, skin, general appearance and others (thigh, abdomen unobtrusive scar, breast, cardio-vascular, constitutional, face, genitalia, genitourinary, gastrointestinal, hematologic, left ankle unobtrusive scar, lymph nodes, lymphatic, malaise/fatigue, mouth, musculoskeletal, musculoskeletal, peripherally inserted central catheters line site left arm, psychiatric, skeletal, urinary, weight, activity level, bladder irritation, dyspnea and eastern cooperative oncology group performance status [used to assess how the disease affects the daily living abilities of the participant. It ranges on the scale from 0-5 (0= normal activity; 1= symptoms but ambulatory; 2= in bed for less than (<) 50 percent (%) of the time; 3= in bed for greater than (>) 50% of the time; 4= 100% bedridden; 5= dead]). Abnormality in physical examinations was based on investigator's discretion.
Time Frame: Baseline (Day 1), Week 1, 4, 8, 12, 24, 36, 48, 52
Population: Safety population included all participants who received at least 1 treatment with dalteparin sodium. Here 'n' signifies those participants who were evaluable at specified categories.
Measure: Number; unit: participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
participants
  Baseline : Head (n=327) | 14
  Baseline : Ears, nose, throat (ENT)(n=327) | 20
  Baseline : Neck (n=327) | 10
  Baseline : Heart (n=327) | 26
  Baseline : Chest (n=326) | 40
  Baseline : Lungs (n=327) | 65
  Baseline : Abdomen (n=327) | 73
  Baseline : Extremities (n=328) | 203
  Baseline : Neurological systems (n=327) | 18
  Baseline : Skin (n=327) | 51
  Baseline : General appearance (n=327) | 47
  Baseline : Others (n=47) | 25
  Week 1 : Head (n=213) | 16
  Week 1 : ENT (n=214) | 20
  Week 1 : Neck (n=214) | 7
  Week 1 : Heart (n=214) | 10
  Week 1 : Chest (n=213) | 22
  Week 1 : Lungs (n=214) | 28
  Week 1 :Abdomen (n=214) | 62
  Week 1 : Extremities (n=213) | 103
  Week 1 : Neurological systems (n=213) | 16
  Week 1 : Skin (n=213) | 52
  Week 1 : General appearance (n=212) | 25
  Week 1:Others (n=41) | 23
  Week 4 : Head (n=211) | 12
  Week 4 : ENT (n=211) | 16
  Week 4 : Neck (n=211) | 6
  Week 4 : Heart (n=210) | 8
  Week 4 : Chest (n=211) | 23
  Week 4 : Lungs (n=211) | 24
  Week 4 : Abdomen (n=210) | 59
  Week 4 : Extremities (n=211) | 83
  Week 4 : Neurological systems (n=211) | 9
  Week 4 : Skin (n=210) | 49
  Week 4 : General appearance (n=208) | 25
  Week 4 : Others (n=23) | 20
  Week 8 : Head (n=186) | 11
  Week 8 : ENT (n=186) | 16
  Week 8 : Neck (n=185) | 4
  Week 8 : Heart (n=186) | 8
  Week 8 : Chest (n=186) | 21
  Week 8 : Lungs (n=186) | 31
  Week 8 : Abdomen (n=186) | 49
  Week 8 : Extremities (n=186) | 80
  Week 8 : Neurological systems (n=185) | 13
  Week 8 : Skin (n=186) | 38
  Week 8 : General appearance (n=186) | 16
  Week 8 : Others (n=16) | 12
  Week 12 : Head (n=183) | 10
  Week 12 : ENT (n=183) | 12
  Week 12 : Neck (n=183) | 1
  Week 12 : Heart (n=183) | 9
  Week 12 : Chest (n=183) | 22
  Week 12 : Lungs (n=183) | 15
  Week 12 : Abdomen (n=183) | 47
  Week 12 : Extremities (n=183) | 57
  Week 12 : Neurological systems (n=183) | 19
  Week 12 : Skin (n=183) | 39
  Week 12 : General appearance (n=182) | 18
  Week 12 : Other (n=27) | 16
  Week 24 : Head (n=166) | 2
  Week 24 : ENT (n=166) | 12
  Week 24 : Neck (n=166) | 4
  Week 24 : Heart (n=166) | 9
  Week 24 : Chest (n=166) | 17
  Week 24 : Lungs (n=166) | 14
  Week 24 : Abdomen (n=166) | 37
  Week 24 : Extremities (n=166) | 47
  Week 24 : Neurological systems (n=166) | 14
  Week 24 : Skin (n=166) | 35
  Week 24 : General appearance (n=166) | 9
  Week 24 : Others (n=17) | 11
  Week 36 : Head (n=127) | 6
  Week 36 : ENT (n=127) | 9
  Week 36 : Neck (n=127) | 4
  Week 36 : Heart (n=127) | 7
  Week 36 : Chest (n=127) | 18
  Week 36 : Lungs (n=127) | 12
  Week 36 : Abdomen (n=126) | 35
  Week 36 : Extremities (n=127) | 37
  Week 36 : Neurological systems (n=127) | 9
  Week 36 : Skin (n=127) | 32
  Week 36 : General appearance (n=126) | 11
  Week 36 : Others (n=14) | 9
  Week 48 : Head (n=103) | 2
  Week 48 : ENT (n=103) | 6
  Week 48 : Neck (n=103) | 3
  Week 48 : Heart (n=103) | 7
  Week 48 : Chest (n=103) | 11
  Week 48 : Lungs (n=102) | 14
  Week 48 : Abdomen (n=103) | 27
  Week 48 : Extremities (n=103) | 29
  Week 48 : Neurological systems (n=103) | 8
  Week 48 : Skin (n=103) | 29
  Week 48 : General appearance (n=103) | 9
  Week 48 : Others (n=7) | 3
  Week 52 : Head (n=193) | 7
  Week 52 : ENT (n=193) | 13
  Week 52 : Neck (n=193) | 5
  Week 52 : Heart (n=193) | 12
  Week 52 : Chest (n=193) | 23
  Week 52 : Lungs (n=191) | 23
  Week 52 : Abdomen (n=193) | 60
  Week 52 : Extremities (n=193) | 68
  Week 52 : Neurological systems (n=193) | 24
  Week 52 : Skin (n=193) | 38
  Week 52 : General appearance (n=193) | 27
  Week 52 : Others (n=25) | 15

17. Other Pre Specified Outcome: Other Pre-specified: Number of Participants With Clinically Significant Electrocardiogram Findings
Description: Clinically significant ECG findings included: corrected QT (QTc) > 450 ms, QTc >500 ms, change in QTc between 30 and 60 ms, change in QTc greater than or equal to 60 ms.
Time Frame: Baseline up to Week 52
Population: Safety population included all participants who received at least 1 treatment with dalteparin sodium.
Measure: Number; unit: participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 334
participants | 8

18. Other Pre Specified Outcome: Change From Baseline in Creatinine Clearance at Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 in Severely Renal Impaired Participants
Description: Creatinine clearance is an indicator of renal function. Creatinine clearance is the volume of blood plasma that is cleared of creatinine by the kidneys per unit time. Normal values for healthy, young males are in the range of 100-135 milliliters per minute (mL/min) and for females, 90-125 mL/min. Creatinine clearance decreases with age.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: Severely renal-impaired population included all participants who had at least 1 dose of study drug and had severe renal impairment at the baseline or developed severe renal impairment (CrCl) < 30 milliliter per minute during the study. Here, n' signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 19
mL/min
  Baseline (n=17) | 46.0 (28.66)
  Week 4 (n=15) | -8.6 (25.39)
  Week 8 (n=13) | 2.5 (47.02)
  Week 12 (n=13) | 2.1 (58.15)
  Week 16 (n=4) | -9.2 (21.93)
  Week 20 (n=2) | 7.7 (7.90)
  Week 24 (n=12) | 4.5 (49.62)
  Week 28 (n=1) | -44.0 (NA) — Standard deviation was not calculated since only 1 participant was evaluable at the given time point.
  Week 32 (n=1) | -14.0 (NA) — Standard deviation was not calculated since only 1 participant was evaluable at the given time point.
  Week 36 (n=8) | 5.8 (56.91)
  Week 40 (n=2) | -21.0 (9.90)
  Week 44 (n=2) | -20.0 (4.24)
  Week 48 (n=6) | -26.0 (18.12)
  Week 52 (n=11) | 4.8 (50.19)

ADVERSE EVENTS:
Arm/Group | Dalteparin Sodium
Serious Adverse Events (participants affected / at risk) | 213/334
Other Adverse Events (participants affected / at risk) | 328/334
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin Sodium (N=334)
Anaemia (Blood and lymphatic system disorders) | 6
Bone marrow failure (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 12
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 4
Pancytopenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Endocarditis noninfective (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Adrenal haemorrhage (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 5
Colitis (Gastrointestinal disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Duodenal obstruction (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Gastrointestinal necrosis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 3
Intestinal perforation (Gastrointestinal disorders) | 2
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Narcotic bowel syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Oesophageal obstruction (Gastrointestinal disorders) | 1
Pancreatic mass (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 3
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 5
Subileus (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Varicose veins of abdominal wall (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Device malfunction (General disorders) | 1
Device occlusion (General disorders) | 2
Disease progression (General disorders) | 29
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 1
Mucosal inflammation (General disorders) | 2
Multi-organ failure (General disorders) | 2
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 2
Pyrexia (General disorders) | 5
Bile duct obstruction (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Cholestasis (Hepatobiliary disorders) | 1
Gallbladder disorder (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bacterial sepsis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Candiduria (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 12
Clostridial infection (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Haematoma infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 2
Lung abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 2
Postoperative wound infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 7
Septic shock (Infections and infestations) | 4
Streptococcal sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 5
Urosepsis (Infections and infestations) | 3
Wound infection (Infections and infestations) | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Inadequate analgesia (Injury, poisoning and procedural complications) | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Procedural complication (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Haemoglobin decreased (Investigations) | 3
Staphylococcus test positive (Investigations) | 1
Weight decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hypovolaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Malignant ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain oedema (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 3
Embolic cerebral infarction (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 2
Haemorrhagic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Stupor (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Thrombotic stroke (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 4
Substance-induced psychotic disorder (Psychiatric disorders) | 1
Calculus bladder (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 4
Postrenal failure (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 5
Renal failure acute (Renal and urinary disorders) | 4
Renal impairment (Renal and urinary disorders) | 1
Ovarian mass (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 20
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 8
Embolism venous (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 4
Jugular vein thrombosis (Vascular disorders) | 1
Subclavian artery stenosis (Vascular disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin Sodium (N=334)
Injection site hematoma (General disorders) | 91
Fatigue (General disorders) | 90
Nausea (Gastrointestinal disorders) | 81
Odema peripheral (General disorders) | 80
Constipation (Gastrointestinal disorders) | 71
Diarrhea (Gastrointestinal disorders) | 60
Anemia (Blood and lymphatic system disorders) | 54
Contusion (Injury, poisoning and procedural complications) | 52
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 52
Decreased appetite (Metabolism and nutrition disorders) | 48
Back pain (Musculoskeletal and connective tissue disorders) | 45
Thrombocytopenia (Blood and lymphatic system disorders) | 42
Vomiting (Gastrointestinal disorders) | 42
Abdominal pain (Gastrointestinal disorders) | 41
Disease progression (General disorders) | 37
Cough (Respiratory, thoracic and mediastinal disorders) | 36
Hypokalemia (Metabolism and nutrition disorders) | 36
Weight decreased (Investigations) | 36
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 34
Pneumonia (Infections and infestations) | 34
Headache (Nervous system disorders) | 33
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33
Urinary tract infection (Infections and infestations) | 32
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 31
Anxiety (Psychiatric disorders) | 27
Dizziness (Nervous system disorders) | 27
Insomnia (Psychiatric disorders) | 27
Neutropenia (Blood and lymphatic system disorders) | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Dehydration (Metabolism and nutrition disorders) | 24
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 24
Pyrexia (General disorders) | 24
Hypotension (Vascular disorders) | 23
Alopecia (Skin and subcutaneous tissue disorders) | 22
Ascites (Gastrointestinal disorders) | 22
Hematuria (Renal and urinary disorders) | 22
Neuropathy peripheral (Nervous system disorders) | 22
Rash (Skin and subcutaneous tissue disorders) | 22
Upper respiratory tract infection (Infections and infestations) | 22
Hyponatremia (Metabolism and nutrition disorders) | 20
Asthenia (General disorders) | 19
Cellulitis (Infections and infestations) | 19
Dry skin (Skin and subcutaneous tissue disorders) | 18
Ecchymosis (Skin and subcutaneous tissue disorders) | 18
Tachycardia (Cardiac disorders) | 18
Hemoglobin decreased (Investigations) | 17
Injection site hemorrhage (General disorders) | 17
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.